CLINICAL TRIAL: NCT06322173
Title: Molecular Diagnostics of Bacterial Infections and Antibiotic Resistance in Blood Samples and Rectal Swabs Using Advanced NGS Sequencing Methods
Acronym: ARES_NGS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Sacro Cuore Don Calabria di Negrar (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022-13
Record Dates: First submitted 2024-03-06; First posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Resistance Bacterial

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NGS analysis (Other): Residual anonymized samples stored at -80°C at the Tropica Biobank of the DITM and for which diagnostic analysis for germ infection has previously been carried out at the DITM by blood culture and MDR surveillance in routine diagnostic rectal swab will be used. DNA extraction will be carried out on these residual samples (with subsequent quality and quantification analysis of the nucleic acid) for subsequent NGS analyses.
  Interventions: Diagnostic Test: NGS Analysis

INTERVENTIONS:
Diagnostic Test: NGS Analysis — An analytical pipeline with NGS technology developed in the GENRES study will be used for the identification of infecting microorganisms and the drug resistance they carry. For this purpose, a sequencing method will be identified and adopted that can obtain gene sequences of approximately 75 bp in length and on the Illumina MiSeq platform. Furthermore, IT software and bioinformatics analyzes with specific quality control parameters (pre- and post-alignment of reads) will be identified and adopted in order to develop an IVD system that includes a complete package of sequencing kits and software.

SUMMARY:
This is an experimental study without drug and device, non-profit, on biological samples stored at the Tropica Biobank of the DITM. The aim of the project is to verify the performance of NGS-based assays, which can be used in the field of microbiology. The clinical evaluation investigations of NGS technology will be conducted on an adequate number of clinical blood samples and rectal swabs. The analyzes will be compared with the standard microbiology methods used in the DITM diagnostic routine.

ELIGIBILITY:
Inclusion criteria:

* Samples of patients for whom blood culture and Multi Drug Resistant (MDR) surveillance tests were carried out in rectal swabs at the IRCCS Sacro Cuore Don Calabria Hospital
* Samples for which the Information and consent to the conservation of biological samples for research purposes has been signed at the Tropica Biobank or
* Samples for which, after all reasonable efforts, it was not possible to obtain the signature of the Information and consent to the conservation of biological samples for research purposes at the Tropica Biobank (e.g. patients in intensive care, immobilized patients unable to sign or with serious alterations of consciousness).

Exclusion criteria:

* Absence of data relating to positivity or negativity to the germs of interest
* Absence of stored residual material

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-06-28 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Microorganism presence (positive/negative) | Baseline
  Microorganism presence identified by NGS technology.
Microorganism identification | Baseline
  Microorganism identification obtained using NGS technology.

SECONDARY OUTCOMES:
Identification of Gene mutations that convey resistance to antibiotics (resistant/susceptible) | Baseline
  Results (resistant/susceptible) obtained using NGS technology in the identification of gene mutations that convey resistance to antibiotics.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Sacro Cuore Don Calabria hospital, Negrar, Verona, Italy